CLINICAL TRIAL: NCT04259840
Title: Clinical Outcomes of Resective Surgical Treatment of Peri-Implantitis With or Without Implantoplasty. A Retrospective Study
Brief Title: Clinical Outcomes of Resective Surgical Treatment of Peri-Implantitis With or Without Implantoplasty
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Collegiate Professor of Periodontics and Professor of Dentistry, University of Michigan
Other Study IDs: HUM00169996
Record Dates: First submitted 2020-01-23; First posted 2020-02-07 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peri-implantitis: Patients who underwent resective surgical treatment for peri-implantitis at the University of Michigan Graduate Periodontics clinic from January 1, 1990 through July 1, 2018
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Soft tissue implant measurements

SUMMARY:
The aims of the current study are 1) to assess the therapeutic resolution of the peri-implantitis after resective surgical treatment with or without implantoplasty procedure (no further radiographic bone loss, no erythema of the peri-implant mucosa, PD <6mm), and 2) to evaluate the survival rate of the peri-implantitis treated dental implants.

DETAILED DESCRIPTION:
The records of patients who underwent resective surgical treatment for peri-implantitis at the University of Michigan Graduate Periodontics clinic will be examined and analyzed. Patients who meet the inclusion/exclusion criteria will be contacted and invited to participate in the study to measure the following in a single visit: bleeding on probing, edema, redness of the peri-implant mucosa, and peri-implant probing pocket depth. Additionally, patients will be asked to complete a survey during their study visit regarding their implant(s) and previous peri-implantitis.

ELIGIBILITY:
Inclusion criteria:

1. The patient is at least 18 years of age,
2. was initially diagnosed with peri-implantitis at ≥1 implant (peri-implant probing depth (PPD) ≥ 6 mm together with bleeding and/or suppuration on probing (BOP/SoP) and bone loss progression over physiological bone remodeling radiologically assessed or marginal bone loss ≥ 3 mm radiologically assessed in case of absence of baseline radiographs),
3. had received treatment for peri-implantitis at least 1 year ago at the Graduate Clinic of Periodontics at University of Michigan, and
4. documentation from ≥ 1 year of clinical and radiological follow- up is available from U of M patients records.

Exclusion criteria:

1. Has received or is currently receiving radiotherapy,
2. are currently pregnant, unsure of their pregnancy status, or are lactating (as reported by the patient),
3. has health condition(s) or takes medication(s) that are known to affect soft tissue or bone (e.g., Phenytoin)
4. Received any kind of bone graft during the treatment of the peri-implantitis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent resective surgical treatment for peri-implantitis at the University of Michigan Graduate Periodontics clinic from January 1, 1990 through July 1, 2018
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Therapeutic resolution of the peri-implantitis as measured by radiographic bone loss | Up to 30 years after the implant was treated for peri-implantitis
  The implant has no further radiographic bone loss when compared to previous radiographs.
Therapeutic resolution of the peri-implantitis as measured by erythema | Up to 30 years after the implant was treated for peri-implantitis
  The implant has no current erythema of the peri-implant mucosa.
Therapeutic resolution of the peri-implantitis as measured by probing depths | Up to 30 years after the implant was treated for peri-implantitis
  The implant has probing depths less than or equal to 5 millimeters.
Survival rate of the peri-implantitis treated dental implants | Up to 30 years after the implant was treated for peri-implantitis
  Survival rate will be determined by the duration of implant survival (functioning, non-symptomatic implant after peri-implantitis treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS MSD PhD, Principal Investigator — Department of Periodontics and Oral Medicine, University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S313-S318. doi: 10.1002/JPER.17-0739. PMID 29926955
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Englezos E, Cosyn J, Koole S, Jacquet W, De Bruyn H. Resective Treatment of Peri-implantitis: Clinical and Radiographic Outcomes After 2 Years. Int J Periodontics Restorative Dent. 2018 Sep/Oct;38(5):729-735. doi: 10.11607/prd.3386. PMID 30113610
- [Background] Hammerle CHF, Tarnow D. The etiology of hard- and soft-tissue deficiencies at dental implants: A narrative review. J Clin Periodontol. 2018 Jun;45 Suppl 20:S267-S277. doi: 10.1111/jcpe.12955. PMID 29926502
- [Background] Heitz-Mayfield LJ. Peri-implant diseases: diagnosis and risk indicators. J Clin Periodontol. 2008 Sep;35(8 Suppl):292-304. doi: 10.1111/j.1600-051X.2008.01275.x. PMID 18724857
- [Background] Khoury F, Buchmann R. Surgical therapy of peri-implant disease: a 3-year follow-up study of cases treated with 3 different techniques of bone regeneration. J Periodontol. 2001 Nov;72(11):1498-508. doi: 10.1902/jop.2001.72.11.1498. PMID 11759861
- [Background] Machtei EE. Treatment Alternatives to Negotiate Peri-Implantitis. Adv Med. 2014;2014:487903. doi: 10.1155/2014/487903. Epub 2014 Jun 15. PMID 26556414
- [Background] Monje A, Blasi G. Significance of keratinized mucosa/gingiva on peri-implant and adjacent periodontal conditions in erratic maintenance compliers. J Periodontol. 2019 May;90(5):445-453. doi: 10.1002/JPER.18-0471. Epub 2018 Dec 7. PMID 30461016
- [Background] Monje A, Galindo-Moreno P, Tozum TF, Suarez-Lopez del Amo F, Wang HL. Into the Paradigm of Local Factors as Contributors for Peri-implant Disease: Short Communication. Int J Oral Maxillofac Implants. 2016 Mar-Apr;31(2):288-92. doi: 10.11607/jomi.4265. PMID 27004275
- [Background] Monje A, Pons R, Insua A, Nart J, Wang HL, Schwarz F. Morphology and severity of peri-implantitis bone defects. Clin Implant Dent Relat Res. 2019 Aug;21(4):635-643. doi: 10.1111/cid.12791. Epub 2019 May 14. PMID 31087457
- [Background] Monje A, Wang HL, Nart J. Association of Preventive Maintenance Therapy Compliance and Peri-Implant Diseases: A Cross-Sectional Study. J Periodontol. 2017 Oct;88(10):1030-1041. doi: 10.1902/jop.2017.170135. Epub 2017 May 26. PMID 28548886
- [Background] Renvert S, Polyzois I, Claffey N. Surgical therapy for the control of peri-implantitis. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:84-94. doi: 10.1111/j.1600-0501.2012.02554.x. PMID 23062132
- [Background] Rimondini L, Fare S, Brambilla E, Felloni A, Consonni C, Brossa F, Carrassi A. The effect of surface roughness on early in vivo plaque colonization on titanium. J Periodontol. 1997 Jun;68(6):556-62. doi: 10.1902/jop.1997.68.6.556. PMID 9203099
- [Background] Roccuzzo M, De Angelis N, Bonino L, Aglietta M. Ten-year results of a three-arm prospective cohort study on implants in periodontally compromised patients. Part 1: implant loss and radiographic bone loss. Clin Oral Implants Res. 2010 May;21(5):490-6. doi: 10.1111/j.1600-0501.2009.01886.x. Epub 2010 Mar 11. PMID 20337668
- [Background] Romeo E, Ghisolfi M, Murgolo N, Chiapasco M, Lops D, Vogel G. Therapy of peri-implantitis with resective surgery. A 3-year clinical trial on rough screw-shaped oral implants. Part I: clinical outcome. Clin Oral Implants Res. 2005 Feb;16(1):9-18. doi: 10.1111/j.1600-0501.2004.01084.x. PMID 15642026
- [Background] Romeo E, Lops D, Chiapasco M, Ghisolfi M, Vogel G. Therapy of peri-implantitis with resective surgery. A 3-year clinical trial on rough screw-shaped oral implants. Part II: radiographic outcome. Clin Oral Implants Res. 2007 Apr;18(2):179-87. doi: 10.1111/j.1600-0501.2006.01318.x. PMID 17348882
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Periodontol. 2018 Jun;89 Suppl 1:S267-S290. doi: 10.1002/JPER.16-0350. PMID 29926957
- [Background] Schwarz F, Sahm N, Becker J. Combined surgical therapy of advanced peri-implantitis lesions with concomitant soft tissue volume augmentation. A case series. Clin Oral Implants Res. 2014 Jan;25(1):132-6. doi: 10.1111/clr.12103. Epub 2013 Jan 27. PMID 23350647
- [Background] Schwarz F, Sahm N, Schwarz K, Becker J. Impact of defect configuration on the clinical outcome following surgical regenerative therapy of peri-implantitis. J Clin Periodontol. 2010 May;37(5):449-55. doi: 10.1111/j.1600-051X.2010.01540.x. Epub 2010 Mar 24. PMID 20374416
- [Background] Zitzmann NU, Berglundh T. Definition and prevalence of peri-implant diseases. J Clin Periodontol. 2008 Sep;35(8 Suppl):286-91. doi: 10.1111/j.1600-051X.2008.01274.x. PMID 18724856
- [Derived] Ravida A, Siqueira R, Saleh I, Saleh MHA, Giannobile A, Wang HL. Lack of Clinical Benefit of Implantoplasty to Improve Implant Survival Rate. J Dent Res. 2020 Nov;99(12):1348-1355. doi: 10.1177/0022034520944158. Epub 2020 Jul 27. PMID 32718212